CLINICAL TRIAL: NCT00294437
Title: Randomised Open-label Multicenter Prosp. Clinical Study to Show the Efficacy of IV ZOMETA® 4mg for Prevention of Bone Metastases in Hormone-naïve High Risk Patients With Locally Advanced Prostate Cancer
Brief Title: ZOMETA® (Zoledronic Acid) for Prevention of Bone Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: underfunding
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: CECOG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/prostate 1.2.001
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Zometa
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- zoledronic acid (Experimental): Zometa® (zoledronic acid) in 100ml of calcium free solution i.v. as a 15 minute infusion every 3 months
  Interventions: Drug: Zometa
- no intervention (No Intervention): no reference therapy

INTERVENTIONS:
Drug: Zometa — Zometa® (zoledronic acid) in 100ml of calcium free solution i.v. as a 15 minute infusion every 3 months
  Arms: zoledronic acid

SUMMARY:
To determine if therapy with Zometa® (zoledronic acid) 4mg will be effective in preventing the occurrence of bone metastases in prostate cancer patients at high risk of developing them. In addition, pain and analgesic scores and overall safety are to be evaluated throughout the study.

DETAILED DESCRIPTION:
This is a prospective, randomized, stratified open-label (Zometa + hormonal ablation versus hormonal ablation alone) multicenter clinical study evaluating the efficacy of Zometa 4mg given every 3 month as an adjunct to hormonal or surgical castration for prevention of bone metastases in locally advanced, high risk prostate cancer patients, who are hormone-naiv at time of randomization. the primary efficacy variable is the time to occurrence of first bone metastases.

Zometa® (zoledronic acid) provided as 4mg lyophilised powder Supplementation 500mg Calcium +400-500IU Vitamin D p.o. qd

Arm A:

Zometa® (zoledronic acid) in 100ml of calcium free solution i.v. as a 15 minute infusion every 3 months

Arm B:

no reference therapy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years
* Histologically confirmed diagnosis of carcinoma of the prostate
* ECOG performance status of 0, 1, or 2
* No radiological evident bone metastasis (negative bone scan or verification of suspected foci as benign lesions by additional radiological examination)
* T3-4 AND highest pre-study PSA >20 ng/ml AND Gleason score = 8 (or Gleason grade = 4)
* Patients with prior prostatectomy or prior local radiotherapy are eligible for this study
* Patients are destined to receive medical (LHRH analogue) or surgical (orchiectomy) castration and Zometa® treatment will start not later than 6 weeks after surgery
* Patients should be fully recovered from prior interventions where applicable

Exclusion Criteria:

* Patients with a serum creatinine determination >265 µmol/L (3.0 mg/dL)
* Patients that received prior medical (LHRH analogue) castration
* Current (or previous) evidence of metastatic disease to the bone
* History of any other neoplasm within the past five years except for nonmelanomatous skin cancer.
* Previous hormonal therapy with LHRH agonists or other forms of hormonal ablation
* WBC<3.0x109, ANC < 1500/mm3, Hgb<8.0 g/dL, platelets < 75 x 109/L
* Liver function tests >2.5 ULN
* Prior treatment with Zometa® (zoledronic acid) or other bisphosphonates
* Treatment with calcitonin, mithramycin, or gallium nitrate within 2 weeks prior to the date of randomization (Visit 2)
* Use of other investigational drugs (drugs not marketed for any indication) within 30 days prior to the date of randomization (Visit 2)
* Patients with evidence in the six months prior to randomization of severe cardiovascular disease (defined as uncontrolled congestive heart failure), hypertension refractory to treatment, or symptomatic coronary artery disease uncontrolled by treatment
* History of noncompliance to medical regimens and patients who are considered potentially unreliable or incapable of giving informed consent as judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2003-12; Primary Completion 2003-12 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Time to occurrence of first bone metastasis, as assessed by bone scan and confirmed by additional radiological examination

SECONDARY OUTCOMES:
To assess the effects of i.v. Zometa® (zoledronic acid) 4 mg, with respect to the following efficacy parameters as well as safety and tolerability:
Effects on pain and analgesic drug consumption, assessed by the composite pain score from BPI (Brief Pain Inventory) for pain and by analgesic score
Time to first event of bone pain
Time to first occurrence of Skeletal Related Events (SREs), defined as pathologic bone fractures, spinal cord compression, surgery to bone, radiation therapy to bone (including the use of radioisotopes)
Proportion of patients in each arm having SRE
Serum PSA
Overall safety

CONTACTS AND LOCATIONS:
Overall Officials: Bobak Djavan, Prof, Principal Investigator — Univ. Klinik für Urologie
Locations (56):
- Austria (7):
  - LKH Leoben, Abt. für Innere Medizin, Leoben, Styria
  - Thermenkh Baden, Urologie, Baden
  - LKH Graz Univ. Klinik f Urologie, Graz
  - LKH Innsbruck, Dept f. Urologie, Innsbruck
  - KH d Elisabethinen Linz, Dep of Urology, Linz
  - KH der Barmherzigen Schwestern, Dept Urologie, Linz
  - LKH Salzburg, Clinic f Radiotherapy a Radiooncology, Salzburg
- Institute for Oncology, Sarajevo, Bosnia and Herzegovina
- Bulgaria (6):
  - Plovdiv Cancer Center, Plovdiv
  - SBALO National Oncology Center, Sofia
  - Sofia Cancer Center compl. Mladost ,, Sofia
  - MODOSZ Oncology Dispensary, Stara Zagora
  - Oncological Hospital, Varna
  - Modozs-Veliko, Veliko Tarnovo
- Croatia (3):
  - Univ. Hospital, Dep of Pathophysiology, Split
  - GH, Dep Oncology and Reumatology, Varaždin
  - Clinical Hospital, Zagreb
- Czechia (4):
  - FH, Urological Clinic, Brno
  - Hospital Kromeriz, Dep of Urology, Kroměříž
  - FN Motol, Dep of Urology, Prague
  - Centre of Oncology, Ústí nad Labem
- Estonia (2):
  - Mustamae Korpus, Tallinn
  - Clinic of surgery, Tartu
- Hungary (5):
  - Dept. Of Urology , Jahn Ferenc Delpesti Hospital, Budapest
  - karolyi sandor Hospital, Dept of Urology, Budapest
  - Semmelweiss Univ of Medicine, Clinic of Urology, Budapest
  - Univ. of Pecs,Urologic Clinic, Pécs
  - Dept. Of Urology and Surgery, Szombathely
- Lithuanian Oncology Center, Vilnius, Lithuania
- Clinical Center of Montenegro, Podgorica, Montenegro
- Poland (4):
  - Centrum Onkologii Instytut, Krakow
  - Medical Academy, Szczecin
  - Central Rail Hospital,, Warsaw
  - Medical Academy, Warsaw
- Romania (6):
  - P.D.R. Clinic, Brasov
  - Fundeni Hospital, Dep of Urology, Bucharest
  - Saint John Emergency Clinical Hospital, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Emergency Clinical County Hospital , Clin Oncol. Dep, Craiova
  - University Hospital, Iași
- Russia (2):
  - Hertzen Research Oncological Institute, Moscow
  - Medical Radiological Research Center, Obninsk
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Oncology Institute Belgrade, Belgrade
  - Oncology Institute, Belgrade
  - Institute for Oncology, Kamenitz
  - Clinical Center, Niš
- Slovakia (3):
  - FNsP - akad L. Derea Urology, Bratislava
  - FNsP Dep of Urology, Košice
  - FN sP Dep of Urology, Martin
- Slovenia (2):
  - University Clinical Center, Ljubljana
  - Gh, Dep of Urology, Maribor
- South Africa (4):
  - Turret House, Claremont
  - Johannesburg Hospital Dep of Urology, Johannesburg
  - St. Annes Hospital, Pietermaritzburg
  - Urological Hospital, Pretoria

REFERENCES:
- See also: Related Info — http://www.cecog.org